CLINICAL TRIAL: NCT07331441
Title: External Oblique Intercostal Plane Block for Postoperative Analgesia After Major Upper Abdominal Surgery: A Randomized Controlled Trial
Brief Title: External Oblique Intercostal Plane Block for Postoperative Analgesia After Major Upper Abdominal Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jun Zhang (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, Department of Anesthesiology of Shanghai cancer center, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2512335-12
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Abdominal Surgery; Postoperative Pain
Keywords: External Oblique Intercostal Plane Block; Postoperative Pain; Laparoscopic Surgery; Pain Management; Randomized Controlled Trial
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EOIB Block (Experimental): Participants receive ultrasound-guided bilateral External Oblique Intercostal Plane Block (EOIB) after induction of general anesthesia and before surgical incision, using ropivacaine (15 mL per side), in addition to standard multimodal analgesia (including IV PCA and ERAS-based non-opioid analgesics).
  Interventions: Procedure: External Oblique Intercostal Plane Block
- Usual Analgesia (Sham Comparator): Participants receive standard multimodal analgesia without any regional block. Analgesia includes IV patient-controlled analgesia (PCA) and other non-opioid analgesics per the institutional ERAS protocol.
  Interventions: Other: Standard multimodal analgesia

INTERVENTIONS:
Procedure: External Oblique Intercostal Plane Block — Ultrasound-guided bilateral external oblique intercostal plane block (EOIB) performed after induction of general anesthesia and before surgical incision. Using an in-plane technique at the 6th rib level, 15 mL per side of local anesthetic solution (ropivacaine 0.75% diluted with normal saline) is injected between the external oblique muscle and the intercostal muscle. Standard multimodal analgesia is also provided to all participants.
  Other Names: EOIB
  Arms: EOIB Block
Other: Standard multimodal analgesia — Standard multimodal analgesia per institutional ERAS practice, including intravenous patient-controlled analgesia (IV PCA) with opioids and adjunct non-opioid analgesics (e.g., NSAIDs and/or acetaminophen) with antiemetic prophylaxis as needed. No regional block is administered.
  Other Names: Usual analgesia
  Arms: Usual Analgesia

SUMMARY:
Postoperative pain after laparoscopic major upper abdominal surgery (e.g., gastric, hepatic, gallbladder, pancreatic surgery) is often severe, and inadequate analgesia may lead to increased opioid use, opioid dependence, and poor functional recovery. Current analgesic techniques such as neuraxial block have safety concerns (e.g., hypotension, neurological injury), while transversus abdominis plane (TAP) block is ineffective for blocking the lateral cutaneous branches of intercostal nerves in the upper abdomen. The External Oblique Intercostal Plane Block (EOIB) is a novel regional block technique that has shown promise in reducing postoperative opioids and pain in small-scale studies, but evidence for its use in major upper abdominal surgery is limited. This randomized controlled trial (RCT) aims to evaluate the analgesic efficacy and safety of bilateral EOIB combined with standard multimodal analgesia versus standard multimodal analgesia alone in patients undergoing elective laparoscopic major upper abdominal surgery. The primary outcome is the total postoperative opioid consumption (measured as Morphine Milligram Equivalents, MME) within 24 hours. Secondary and additional outcomes include pain scores (Verbal Rating Scale, VRS), recovery quality (QoR-15 scale), incidence of adverse events, and hospital stay.

DETAILED DESCRIPTION:
Postoperative pain after major upper abdominal surgery is common and may delay recovery and increase opioid-related adverse effects. The External Oblique Intercostal Plane Block (EOIB) is a novel fascial plane block intended to improve analgesia for upper abdominal incisions.

This study is a prospective, single-center, randomized, assessor-blinded controlled trial in adults (18-85 years, ASA I-III) scheduled for elective major upper abdominal laparoscopic-assisted surgery (e.g., gastric, hepatic, gallbladder, pancreatic procedures) with expected operative time ≥2 hours and planned use of IV patient-controlled analgesia (PCA). Participants will be randomized 1:1 using a computer-generated, variable block-size sequence with allocation concealment via opaque sealed envelopes. The block-performing anesthesiologist will not collect outcomes; outcome assessors will be blinded to group assignment.

After induction of general anesthesia and before surgical incision, patients in the intervention group will receive ultrasound-guided bilateral EOIB at the 6th rib level using an in-plane technique; 15 mL per side of a mixture of 0.75% ropivacaine and normal saline will be injected. Control participants will receive no regional block. All participants will receive standardized multimodal analgesia including IV PCA, antiemetic prophylaxis (dexamethasone 5 mg; ondansetron as needed), and NSAID use per ERAS practice.

The primary endpoint is total opioid consumption during the first 24 hours after surgery, expressed as IV morphine milligram equivalents (MME), including PCA and rescue opioids. Secondary outcomes include postoperative pain scores (0-10 verbal rating scale) at prespecified time points (including 24, 48, and 72 hours; at rest and with activity as applicable), quality of recovery (QoR-15 at 24/48/72 hours), opioid consumption at 24-48 hours, postoperative nausea and vomiting within 72 hours, intraoperative hemodynamic events, time to first flatus, and postoperative length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Obtain written informed consent from participants or their legal representatives
* Age between 18 and 85 years
* American Society of Anesthesiologists (ASA) physical status classification I-III
* Scheduled for elective laparoscopic major upper abdominal surgery (e.g., gastric, hepatic, gallbladder, pancreatic surgery)
* Expected surgical duration ≥ 2 hours
* Ability to use the intravenous patient-controlled analgesia (IV PCA) system

Exclusion Criteria:

* Hepatic disease (liver enzyme levels ≥ 2× the upper limit of normal)
* Renal disease (serum creatinine levels ≥ 2× the upper limit of normal)
* Allergy to local anesthetics or known study-related drugs
* Pregnancy or lactation
* Low surgical incision site (not involving the upper abdominal wall innervated by T6-T10 nerves)
* Coagulopathy or current use of anticoagulant medications
* Opioid use for more than 2 weeks in the past 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Total opioid consumption within 24 hours after surgery (IV morphine milligram equivalents, MME) | 0-24 hours postoperatively (from end of surgery to 24 hours after surgery)
  Cumulative postoperative opioid use from end of surgery to 24 hours postoperatively, including IV PCA opioids and any rescue opioids, converted to intravenous morphine milligram equivalents (MME) and reported in mg.

SECONDARY OUTCOMES:
Postoperative Pain Score Within 24 Hours Postoperatively | Within 24 hours postoperatively
  Pain is assessed using a Verbal Rating Scale (VRS) with scores ranging from 0 (no pain) to 10 (worst pain imaginable). Assessments are performed each morning and evening. A difference of ≥1 point between groups is considered clinically significant.
Postoperative Recovery Quality at 24 Hours Postoperatively | 24 hours postoperatively
  Recovery quality is evaluated using the QoR-15 scale (a 15-item questionnaire measuring physical comfort, emotional state, and functional recovery). A difference of ≥6 points between groups is considered clinically significant.

OTHER OUTCOMES:
Opioid Consumption (Morphine Milligram Equivalents, MME) Within 24-48 Hours Postoperatively | 25-48 hours postoperatively
  Total opioid consumption includes doses from intravenous patient-controlled analgesia (IV PCA) and rescue analgesics, converted to Morphine Milligram Equivalents (MME). A reduction of ≥10 mg MME between groups is considered clinically significant.
Postoperative Pain Score Postoperatively | 25~72 hours postoperatively
  Pain is assessed using a Verbal Rating Scale (VRS) with scores ranging from 0 (no pain) to 10 (worst pain imaginable). Assessments are performed each morning and evening. A difference of ≥1 point between groups is considered clinically significant.
Postoperative Recovery Quality Postoperatively | 25~72 hours postoperatively
  Recovery quality is evaluated using the QoR-15 scale (a 15-item questionnaire measuring physical comfort, emotional state, and functional recovery). A difference of ≥6 points between groups is considered clinically significant.
Incidence of Nausea and Vomiting Postoperatively | Within 72 hours postoperatively (stratified by 1-6h, 7-24h, 25-48h, 49-72h)
  The number of patients experiencing nausea or vomiting is recorded, stratified by four time periods: 1-6 hours, 7-24 hours, 25-48 hours, and 49-72 hours postoperatively.
Intraoperative Incidence of Hypotension and Hypertension | Intraoperatively (during surgery)
  Intraoperative hypotension is defined as systolic blood pressure <90 mmHg or a 30% reduction from baseline; intraoperative hypertension is defined as systolic blood pressure >160 mmHg or a 30% increase from baseline. The incidence of both conditions is recorded.
Time to First Flatus Postoperatively | From surgery completion to first flatus (up to 72 hours postoperatively)
  The duration from surgery completion to the patient's first flatus is recorded as an indicator of gastrointestinal function recovery.
Postoperative Hospital Stay Duration | From surgery completion to hospital discharge (typically 3-7 days postoperatively)
  The duration from surgery completion to hospital discharge is recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, PhD, Study Director — Fudan University

IPD SHARING:
Plan to Share IPD: No